CLINICAL TRIAL: NCT05925296
Title: The Effect of Dual-site Repetitive Transcranial Magnetic Stimulation on Freezing of Gait in Patients With Parkinson Disease
Brief Title: The Effect of Dual-site Repetitive Transcranial Magnetic Stimulation on Freezing of Gait in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kezhong Zhang, Professor/Chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-SRFA-020
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: freezing of gait; rTMS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- double-site high frequency rTMS over the bilateral M1 of the lower leg and SMA (Experimental): Patients in the Experimental group underwent ten sessions of double-site high frequency rTMS over the bilateral M1 of the lower leg and SMA.
  Interventions: Device: magnetic stimulation
- single-site high frequency rTMS over the bilateral primary motor cortex of the lower leg (Active Comparator): Patients in the Active Comparator group underwent ten sessions of single-site active magnetic stimulation with high frequency rTMS over the bilateral M1 of the lower leg.
  Interventions: Device: magnetic stimulation
- sham magnetic stimulation on motor cortex (Sham Comparator): Patients in the Sham Comparator group underwent 10 sessions of double sham rTMS on M1.
  Interventions: Device: magnetic stimulation

INTERVENTIONS:
Device: magnetic stimulation — Patients in the Experimental group underwent ten sessions of double-site high frequency rTMS over the bilateral primary motor cortex of the lower leg and supplementary motor area, whereas patients in the Active Comparator group underwent ten sessions of single-site active magnetic stimulation with high frequency rTMS over the bilateral primary motor cortex of the lower leg. In addition, patients in the Sham Comparator group underwent 10 sessions of double sham rTMS on motor cortex.

SUMMARY:
This study is a double-blinded randomized study examining the effectiveness of the dual-site repetitive transcranial magnetic stimulation on Freezing of Gait (FOG) in patients with Parkinson's disease. The investigators hypothesize that treatment using magnetic stimulation on double site (including M1-LL and SMA) will improve FOG and gait symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Patients in the Experimental group underwent ten sessions of double-site high frequency rTMS over the bilateral primary motor cortex of the lower leg and supplementary motor area, whereas patients in the Active Comparator group underwent ten sessions of single-site active magnetic stimulation with high frequency rTMS over the bilateral primary motor cortex of the lower leg. In addition, patients in the Sham Comparator group underwent 10 sessions of double sham rTMS on motor cortex. Assessments of FOG, gait function, motor symptoms, excitability of cortex motor (using transcranial magnetic stimulation), plasma indicators and multimodal magnetic resonance were performed three times: at baseline, one day post intervention, one month post intervention, six month post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease (PD), as diagnosed by a neurologist.
2. Item 3 of the Freezing of Gait Questionnaire(FOG-Q) scored ≥1.
3. Age between 40 and 80 years old.
4. Mini-Mental State Examination score >24.
5. Ability to walk 30 meters independently.
6. Stable medication.
7. Patients experienced FOG during an interview.

Exclusion Criteria:

1. Other neurological or psychiatric disorders.
2. Severe personality disorder. History of epilepsy, seizures, or convulsions.
3. History of head injury or stroke.
4. Metal remains of the skull or inside the brain (outside the oral cavity).
5. Surgeries including metallic implants or known history of metal particles in the eye, pacemakers,hearing devices transplantation, or medical pumps.
6. Severe dyskinesia, tremor, cognitive, visual or auditory impairment.
7. Patients who could not complete the follow-up.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Freezing of Gait Questionnaire | Assessed at baseline, one day post intervention, one month post intervention, six months post intervention
  The Freezing of Gait questionnaire will be used to quantify the frequency and severity of this symptom. The score will be compared to the baseline. The minimum and maximum values of the FOG-Q are 0 and 24. A higher FOG-Q score means a worse outcome. The differences in FOG-Q scores before and after treatment can be used to evaluate the effect of TMS treatment.

SECONDARY OUTCOMES:
Changes of MDS-UPDRS | Assessed at baseline, one day post intervention, one month post intervention, six months post intervention
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms and non-motor symptoms. A higher score means a worse outcome. The score will be compared to the baseline. The differences in MDS-UPDRS scores before and after treatment can be used to evaluate the effect of TMS treatment.
Gait speed | Assessed at baseline, one day post intervention, one month post intervention, six month post intervention
  Gait speed (m/s) was evaluated at baseline, one day post intervention, one month post intervention, six month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test. The differences in gait speed before and after treatment can be used to evaluate the effect of TMS treatment.
Stride length | Assessed at baseline, one day post intervention, one month post intervention, six month post intervention
  Stride length (cm) was evaluated at baseline, one day post intervention, one month post intervention, six month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test. The differences in stride length before and after treatment can be used to evaluate the effect of TMS treatment.
Stride time variability | Assessed at baseline, one day post intervention, one month post intervention, six month post intervention
  Stride time variability (%) was evaluated at baseline, one day post intervention, one month post intervention, six month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test. The differences in stride time variability before and after treatment can be used to evaluate the effect of TMS treatment.
Double support | Assessed at baseline, one day post intervention, one month post intervention, six month post intervention
  Double support (%) was evaluated at baseline, one day post intervention, one month post intervention, six month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test. The differences in double support before and after treatment can be used to evaluate the effect of TMS treatment.
Resting motor threshold (RMT) | Assessed at baseline, one day post intervention
  RMT (% TMS output intensity) is defined as the lowest intensity required to elicit MEPs of > 50 μV in at least 5 of 10 consecutive trials while the target muscle is relaxed. RMT was determined to be the nearest 1% of the maximum stimulator output. The differences in RMT before and after treatment can be used to evaluate the effect of TMS treatment.
Cortical silent period (CSP) | Assessed at baseline, one day post intervention
  The CSP (ms) is measured through electromyographic signal recording (EMG) on a target muscle and refers to the period of EMG silence following the elicitation of a motor-evoked potential (MEP) through a single TMS pulse delivered over the contralateral primary motor cortex. The differences in CSP before and after treatment can be used to evaluate the effect of TMS treatment.
Short-interval intracortical inhibition (SICI) | Assessed at baseline, one day post intervention
  SICI was assessed with a subthreshold conditioning stimulus (80% RMT) and a supra-threshold test stimulus (1 mV MEP) with 2ms, 3ms, 4ms interstimulus interval between conditioning and test stimuli. Ten trials were acquired for each interstimulus interval. SICI was expressed as the percentage ratio between the test and conditioning MEP. The differences in SICI before and after treatment can be used to evaluate the effect of TMS treatment.
Intracortical facilitation (ICF) | Assessed at baseline, one day post intervention
  ICF was assessed with a subthreshold conditioning stimulus (80% RMT) and a supra-threshold test stimulus (1 mV MEP) with 10ms, 12, 15 ms interstimulus interval between conditioning and test stimuli. Ten trials were acquired for each interstimulus interval. ICF was expressed as the percentage ratio between the test and conditioning MEP. The differences in ICF before and after treatment can be used to evaluate the effect of TMS treatment.
Short-interval intracortical facilitation (SICF) | Assessed at baseline, one day post intervention
  A subthreshold first stimulus (S1) intensity was set at 1 mV and a subsequent suprathreshold second stimulus (S2) intensity was set at RMT. Interstimulus intervals were 1.0 to 5.0 milliseconds with increments of 0.5 millisecond. Ten trials for each and ten single-pulse trials were given in randomized order. SICF was expressed as the percentage ratio between the S1 and S2 MEP. The differences in SICF before and after treatment can be used to evaluate the effect of TMS treatment.
Plasma indicators | Assessed at baseline, one day post intervention
  5ml of the patient's elbow vein blood was collected and centrifuged after standing and stratified. The blood plasma was collected and frozen at - 80°C for testing. Detection of changes in plasma BDNF levels. The differences in BDNF before and after treatment can be used to evaluate the effect of TMS treatment.
Changes in functional connectivity in the brain cortex | Assessed at baseline, one day post intervention, six month post intervention
  The functional connectivity in the brain cortex will be recorded by functional MRI. The differences in brain regions' functional connectivity before and after treatment can be used to evaluate the effect of TMS treatment.
Changes in cerebral blood flow in the brain cortex | Assessed at baseline, one day post intervention, six month post intervention
  The cerebral blood flow will be assessed by arterial spin labeling scanning. The differences in blood flow before and after treatment can be used to evaluate the effect of TMS treatment.
Brian structure compared among groups | Assessed at baseline, one day post intervention, six month post intervention
  Studying the brain structure among groups. The differences in brain microstructure before and after treatment can be used to evaluate the effect of TMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No